CLINICAL TRIAL: NCT02239211
Title: A Single Arm, Two-stage, Multi-centre, Phase II Clinical Trial Investigating the Safety and Activity of the Use of BTT1023 Targeting Vascular Adhesion Protein (VAP-1), in the Treatment of Patients With Primary Sclerosing Cholangitis (PSC).
Brief Title: A Trial of BTT1023 in Patients With Primary Sclerosing Cholangitis
Acronym: BUTEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Biotie Therapies Corp. (Industry); University Hospital Birmingham (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_13-027; 2014-002393-37 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: BUTEO; Primary sclerosing cholangitis; PSC; VAP-1; BTT1023; Human monoclonal antibody
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — timolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BTT1023 (Experimental): BTT1023 8mg/kg IV infusion, total of 7 infusions over 11 weeks. Duration 1-2 hours per infusion.
  Interventions: Drug: BTT1023

INTERVENTIONS:
Drug: BTT1023 — IV (in the vein) Investigational Medicinal Product (IMP)

SUMMARY:
This is a phase II study to determine the safety and preliminary efficacy of a human monoclonal antibody (BTT1023) which targets the vascular adhesion protein (VAP-1) and its use in the treatment of patients with primary sclerosing cholangitis (PSC).

DETAILED DESCRIPTION:
Primary sclerosing cholangitis is a progressive immune mediated biliary disease characterised by bile duct inflammation and fibrosis, and accompanying hepatic fibrosis. For patients with elevated alkaline phosphatase (ALP) in particular, progressive disease is predicted, that currently results in a need for liver transplantation in the majority. No current medical therapy has as yet been shown to be effective in altering the natural history of disease. For this reason patients with PSC with elevated ALP values will be recruited to this study, to evaluate the impact of Vap-1 blockade by BTT1023, in an early phase study focused on biochemical efficacy and safety.

This is an early phase study of BTT1023 in immune mediated liver disease, with the rationale to identify biochemical efficacy of effect (reduction in ALP) and safety, in an orphan disease indication for PSC that presently lacks any other medical therapy. The study design therefore focuses on identifying early biochemical efficacy signals to justify larger scale, randomised controlled studies over longer duration.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 - 75 years of age who are willing and able to provide informed, written consent and comply with all trial requirements
2. Clinical diagnosis of PSC as evident by chronic cholestasis of more than six months duration with either a consistent MRI showing sclerosing cholangitis or a liver biopsy consistent with PSC in the absence of a documented alternative aetiology for sclerosing cholangitis
3. In those with concomitant Inflammatory Bowel Disease, clinical and colonoscopic evidence, (in line with the patient's standard of care; within 18 months) of stable disease, without findings of high grade dysplasia
4. In those on treatment with UDCA, therapy must be stable for at least 3 months, and at a dose not greater than 20 mg/kg/day. In those not on treatment with UDCA at the time of screening, a minimum of 8 weeks since the last dose of UDCA should be recorded
5. Serum ALP greater than 1.5 x ULN
6. Stable serum ALP levels (levels must not change by more than 25% from Screening Visit 1 and Screening Visit 2)
7. Female subjects of childbearing potential must have a negative pregnancy test prior to starting trial treatment. For the purposes of this trial, a female subject of childbearing potential is a woman who has not had a hysterectomy, bilateral oophorectomy, or medically-documented ovarian failure. Women ≤ 50 years of age with amenorrhea of any duration will be considered to be of childbearing potential
8. All sexually active women of childbearing potential must agree to use two forms of highly effective method of contraception from the Screening Visit throughout the trial period and for 99 days following the last dose of trial drug. If using hormonal agents the same method must have been used for at least 1 month before trial dosing and subjects must use a barrier method as the other form of contraception. Lactating women must agree to discontinue breast feeding before trial investigational medicinal product administration
9. Men, if not vasectomised, must agree to use barrier contraception (condom plus spermicide) during heterosexual intercourse from screening through to trial completion and for 99 days from the last dose of trial investigational medicinal product
10. Patients must weigh ≥ 40 kg

Exclusion Criteria:

1. Presence of documented secondary sclerosing cholangitis on prior clinical investigations
2. Presence of alternative causes of liver disease, that are considered by the Investigator to be the predominant active liver injury at the time of screening, including viral hepatitis, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis. Patients with possible overlap syndrome with autoimmune hepatitis are excluded if the Investigator considers autoimmune hepatitis as the predominant liver injury
3. AST and ALT >10 x ULN or bilirubin >3 x ULN or INR >1.3 in the absence of anti-coagulants
4. Serum creatinine >130μmol/L or platelet count <50 x 109/L
5. Any evidence of hepatic decompensation past or present, including ascites, episodes of hepatic encephalopathy or variceal bleeding
6. Recent cholangitis within last 90 days or ongoing need for prophylactic antibiotics
7. Pregnancy or breast feeding
8. Harmful alcohol consumption as evaluated by the Investigator
9. Flare in colitis activity within last 90 days requiring intensification of therapy beyond baseline maintenance treatment; use of oral prednisolone >10 mg/day, biologics (i.e. monoclonal antibodies) and or hospitalisation for colitis within 90 days. Prior use of biologics is not a contraindication to screening
10. Diagnosed cholangiocarcinoma or high clinical suspicion of cholangiocarcinoma either clinically or by imaging
11. Concurrent malignancies or invasive cancers diagnosed within past 3 years except for adequately treated basal cell and squamous cell carcinoma of the skin and in situ carcinoma of the uterine cervix
12. Presence of a percutaneous drain or bile duct stent
13. Major surgical procedure within 30 days of screening
14. Prior organ transplantation
15. Known hypersensitivity to the investigational product or any of its formulation excipients
16. Unavailable for follow-up assessment or concern for subject's compliance
17. Participation in an investigational trial of a drug or device within 60 days of screening or 5 half lives of the last dose of investigational drug, where the trial drug half-life is greater than 12 days
18. Any other condition that in the opinion of the Investigator renders the subject a poor risk for inclusion into the trial
19. Positive screening test for tuberculosis (TB) (including T-SPOT.TB TB test), unless respiratory review confirms false positive test results
20. Receipt of live vaccination within 6 weeks prior to Screening Visit 2
21. Known HIV positive status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Response at Visit 10 (Day 99): a reduction in serum ALP by 25% or more from baseline to Visit 10 (Day 99) | 99 days

SECONDARY OUTCOMES:
Treatment Compliance (including patient withdrawal) | 120 days
  These will be measured to evaluate the tolerability of BTT1203 in patients with PSC
Serious Adverse Event (SAE) frequency | 120 days
  These will be measured to evaluate the safety, effective dose, and tolerability of BTT1203 in patients with PSC
Adverse Event (AE) frequency | 120 days
  These will be measured to evaluate the safety, effective dose, and tolerability of BTT1203 in patients with PSC
Calculation of any change (improvement or worsening) from baseline to Day 99 in the quality of life questionnaire EQ-5D | 99 days
  Using validated EQ-5D scoring system
Calculation of any change (improvement or worsening) from baseline to Day 99 in the quality of life questionnaire Fatigue Severity Scale | 99 days
  The scoring is done by calculating the average response to the questions (adding up all the answers and dividing by nine).
Calculation of any change (improvement or worsening) from baseline to Day 99 in the quality of life questionnaire Pruritus Visual Analogue Score | 99 days
  VAS measured as per guidelines
Calculation of any change (improvement or worsening) from baseline to Day 99 in Inflammatory Bowel Disease Diaries (if applicable) | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in enhanced liver fibrosis test | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Fibroscan measures | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Aspartate Transaminase (AST) | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Alanine Transaminase (ALT) | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Alkaline Phosphatase (ALP) | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Gamma Glutamyl Transferase (GGT) | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Bilirubin | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Albumin | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in International Normalised Ratio (INR) | 99 days
Calculation of any change (improvement or worsening) from baseline to Day 99 in Mayo PSC Risk Score | 99 days
  PSC Risk score calculated as per The Revised Natural History Model for Primary Sclerosing Cholangitis
Calculation of any change (improvement or worsening) from baseline to Day 99 in Model for End Stage Liver Disease (MELD) Score | 99 days
  MELD calculated as per pre 2016 guidelines
Evaluate changes (improvement or worsening) in sVAP-1/SSAO as a biomarker of liver disease activity across the trial period | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Newsome, MD, Principal Investigator — University of Birmingham
Locations (6):
- United Kingdom (6):
  - Queens Medical Centre, Nottingham, Nottinghamshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Addenbrooke's Hospital, Cambridge
  - Royal Free Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arndtz K, Corrigan M, Rowe A, Kirkham A, Barton D, Fox RP, Llewellyn L, Athwal A, Wilkhu M, Chen YY, Weston C, Desai A, Adams DH, Hirschfield GM; BUTEO trial team. Investigating the safety and activity of the use of BTT1023 (Timolumab), in the treatment of patients with primary sclerosing cholangitis (BUTEO): A single-arm, two-stage, open-label, multi-centre, phase II clinical trial protocol. BMJ Open. 2017 Jul 3;7(6):e015081. doi: 10.1136/bmjopen-2016-015081. PMID 28674140